CLINICAL TRIAL: NCT06602258
Title: A Phase 2, Placebo-Controlled, Double-Blind, Parallel-Group, Dose-Finding Study to Evaluate Safety, Tolerability, and Biomarker Efficacy of E2814 With Concurrent Lecanemab Treatment in Subjects With Early Alzheimer's Disease
Brief Title: A Study of E2814 With Concurrent Lecanemab Treatment in Participants With Early Alzheimer's Disease
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E2814-G000-202
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer's Disease
Keywords: Early Alzheimer's Disease; E2814; Lecanemab
MeSH Terms: conditions — Alzheimer Disease | interventions — lecanemab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- E2814 Dose A + Lecanemab (Experimental): Participants will receive E2814 Dose A administered as an intravenous (IV) infusion, every four weeks (Q4W) along with lecanemab administered as a subcutaneous (SC) injection, every week (QW).
  Interventions: Drug: E2814; Drug: Lecanemab
- E2814 Dose B + Lecanemab (Experimental): Participants will receive E2814 Dose B administered as an IV infusion, Q4W along with lecanemab administered as a SC injection, QW.
  Interventions: Drug: E2814; Drug: Lecanemab
- E2814 Dose C + Lecanemab (Experimental): Participants will receive E2814 Dose C administered as an IV infusion, Q4W along with lecanemab administered as a SC injection, QW.
  Interventions: Drug: E2814; Drug: Lecanemab
- E2814 Dose D + Lecanemab (Experimental): Participants will receive E2814 Dose D administered as an IV infusion, Q4W along with lecanemab administered as a SC injection, QW.
  Interventions: Drug: E2814; Drug: Lecanemab
- Placebo + Lecanemab (Experimental): Participants will receive placebo administered as an IV infusion, Q4W along with lecanemab administered as a SC injection, QW.
  Interventions: Drug: Lecanemab; Drug: Placebo

INTERVENTIONS:
Drug: E2814 — E2814 IV infusion.
  Arms: E2814 Dose A + Lecanemab; E2814 Dose B + Lecanemab; E2814 Dose C + Lecanemab; E2814 Dose D + Lecanemab
Drug: Lecanemab — Lecanemab SC injection.
  Other Names: BAN2401; LEQEMBI
Drug: Placebo — Placebo IV infusion.
  Arms: Placebo + Lecanemab

SUMMARY:
The primary objective of the study is to determine the dose response of E2814, when concurrently administered with lecanemab, on the change from baseline at 6 months in cerebrospinal fluid (CSF) microtubule-binding region (MTBR)-tau-243 in participants with early Alzheimer's disease (AD).

ELIGIBILITY:
Inclusion Criteria:

1. For participants diagnosed with mild cognitive impairment (MCI) due to AD-intermediate likelihood:

   1. Meet the National Institute on Aging-Alzheimer's Association (NIA-AA) core clinical criteria for MCI due to AD-intermediate likelihood
   2. Have a global Clinical Dementia Rating Scale (CDR) score of 0.5 and a CDR Memory Box score of greater than or equal to (>=) 0.5 at Screening
2. For participants diagnosed with mild AD dementia:

   1. Meet the NIA-AA core clinical criteria for probable AD dementia
   2. Have a global CDR score of 0.5 to 1.0 and a CDR Memory Box score of >=0.5 at Screening
3. Mini Mental State Examination (MMSE) score >=22 at Screening and less than or equal to (<=) 30 at Screening
4. Able to have CSF lumbar puncture performed and not on, or have a medical condition that may require initiation of, any anticoagulant therapy at Screening
5. Male or female participants aged between >=50 years and <=80 years, at the time of informed consent
6. If receiving an approved AD symptomatic treatment (such as acetylcholinesterase inhibitors (AchEIs), memantine, or both) for AD, participants must be on a stable dose for at least 12 weeks before Baseline. Treatment-naïve participants for AD medications can be enrolled into the study. Unless otherwise stated, participants must have been on stable doses of all other (that is, non AD-related) permitted concomitant medications for at least 4 weeks before Baseline. Use of memantine will not be allowed at screening for participants in Japan
7. Have an identified study partner (defined as a person able to support the participant for the duration of the study and who spends at least 8 hours per week with the participant).
8. Provide written informed consent. If a participant lacks the capacity to consent in the Investigator's opinion, the participants' assent should be obtained, if required in accordance with local laws, regulations, and customs, plus the written informed consent of a legal representative should be obtained (capacity to consent and definition of legal representative should be determined in accordance with applicable local laws and regulations)
9. Willing and able to comply with all aspects of the protocol including multiple CSF collections

Exclusion Criteria:

1. Any neurological condition that may be contributing to cognitive impairment above and beyond that caused by the participant's AD
2. History of transient ischemic attacks, stroke, or seizures within 12 months of Screening
3. Any psychiatric diagnosis or symptoms (example, hallucinations, major depression, or delusions) that could interfere with study procedures in the participants. Psychotic disorder(s) or unstable recurrent affective disorder(s) evident by use of antipsychotics within 2 years before Screening
4. Contraindications to MRI scanning, including cardiac pacemaker/defibrillator, ferromagnetic metal implants (example, in skull and cardiac devices other than those approved as safe for use in MRI scanners). Evidence of other clinically significant lesions on brain MRI at Screening that could indicate a dementia diagnosis other than AD. Other significant pathological findings on brain MRI at Screening, including but not limited to: greater than 4 microhemorrhages (defined as 10 millimeter (mm) or less at the greatest diameter); a single intracerebral hemorrhage greater than 10 mm at greatest diameter; an area of superficial siderosis; evidence of vasogenic edema; evidence of cerebral contusion, encephalomalacia, aneurysms, vascular malformations, or infective lesions; evidence of multiple lacunar infarcts or stroke involving a major vascular territory, severe small vessel, or white matter disease; space occupying lesions; or brain tumors (however, lesions diagnosed as meningiomas or arachnoid cysts and less than 1 cm at their greatest diameter need not be exclusionary). Other minor or clinically insignificant magnetic resonance imaging (MRI) abnormalities, as agreed by the medical monitor and after discussion with the investigator, may not be exclusionary
5. Malignant neoplasms within 3 years of Screening (except for basal or squamous cell carcinoma in situ of the skin, or localized prostate cancer in male participants, or localized breast cancer in female participants). Participants who had malignant neoplasms but who have had at least 3 years of documented uninterrupted remission before Screening need not be excluded
6. A clinically significant ECG abnormality, including a marked prolonged corrected QT interval (Fridericia's Correction Formula; QTcF) interval (example, a repeated demonstration of a QTcF interval greater than (>) 450 milliseconds [ms])
7. Participants with a bleeding disorder that is not under adequate control (including a platelet count <50,000 or international normalized ratio [INR] >1.5). Any participants who are on anticoagulant therapy are not permitted to be enrolled
8. Have thyroid-stimulating hormone above normal range. Other tests of thyroid function with results outside the normal range should only be exclusionary if they are considered clinically significant by the investigator. This applies to all participants whether or not they are taking thyroid supplements
9. Abnormally low serum vitamin B12 levels for the testing laboratory (if participant is taking vitamin B12 injections, level should be at or above the lower limit of normal for the testing laboratory). Levels of vitamin B12 may be confirmed with reflex testing to include methylmalonic acid analysis, if available in region
10. Any suicidal ideation with intent with or without a plan at Screening, Baseline, or within 6 months of Screening (that is, answering "Yes" to questions 4 or 5 on the Suicidal Ideation section of the Columbia-Suicide Severity Rating Scale [C-SSRS]) Type 4 or 5, or any suicidal behavior assessment within 6 months before Screening, at Screening, or at the Baseline Visit, or has been hospitalized or treated for suicidal behavior in the past 5 years before Screening)
11. Evidence of clinically significant disease (example, cardiac, respiratory, gastrointestinal, and renal disease) that in the opinion of the investigator(s) could affect the participants safety or interfere with the study assessments. Any other medical conditions (example, cardiac, respiratory, gastrointestinal, and renal disease) that are not stably and adequately controlled or that in the opinion of the investigator(s) could affect the participant's safety or interfere with the study assessments
12. Hypersensitivity to lecanemab, E2814, or any of the excipients
13. Any immunological disease, that is not adequately controlled, or that requires treatment with immunoglobulins, systemic monoclonal antibodies (mAbs) (or derivatives of mAbs), systemic immunosuppressants, or plasmapheresis during the study
14. Any history of or concomitant medical condition that in the opinion of the investigator(s) would compromise the participant's ability to safely complete the study
15. Planned surgery that requires general, spinal, or epidural anesthesia that would take place during the study. Planned surgery that requires only local anesthesia and that can be undertaken as a day case without inpatient stay postoperatively need not result in exclusion if in the opinion of the investigator this operation does not interfere with study procedures and participant safety
16. Known to be human immunodeficiency virus positive
17. Known or suspected history of drug or alcohol abuse or dependence within 2 years before Screening or a positive urine drug test at Screening. Participants who test positive for benzodiazepines or opioids in urine drug testing need not be excluded if in the clinical opinion of the investigator, this is due to the participant taking prior/concomitant medications containing benzodiazepines or opioids for a medical condition and not due to drug abuse
18. Severe visual or hearing impairment that would prevent the participant from performing psychometric tests accurately
19. Participation in a clinical study involving any antiamyloid plaque lowering or anti-tau therapies (including any mAb and antisense oligonucleotide therapies unless it can be documented that the subject only received placebo)
20. Participation in a clinical study involving any therapeutic mAb, protein derived from a mAb, immunoglobulin therapy, or vaccine within 6 months before Screening unless it can be documented that the subject only received placebo

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-12-03 (Estimated); Study Completion 2027-08-18 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in CSF MTBR-tau-243 at 6 Months | Baseline at 6 months

SECONDARY OUTCOMES:
Change From Baseline in Tau Positron Emission Tomography (PET) up to 24 Months | Baseline up to 24 months
Change From Baseline in Clinical Dementia Rating Scale-Sum of Boxes (CDR-SB) up to 24 Months | Baseline up to 24 months
Change From Baseline in Alzheimers Disease Cooperative Scale-Activities of Daily Living Mild Cognitive Impairment Version (ADCS MCI-ADL) up to 24 Months | Baseline up to 24 months
Serum Anti-E2814 Antibody (ADA) Concentration | Baseline up to 27 months
AUC: Area Under the Serum Concentration Versus Time Curve of E2814 | Baseline up to 27 months
Cav: Average Serum Concentration of E2814 | Baseline up to 27 months
Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | From first dose of the study drug up to 27 months
Number of Participants With Markedly Abnormal Laboratory Parameters | From first dose of the study drug up to 27 months
Number of Participants With Clinically Significant Vital Signs Values | From first dose of the study drug up to 27 months
Number of Participants With Clinically Significant Electrocardiogram (ECG) Findings | From first dose of the study drug up to 27 months

CONTACTS AND LOCATIONS:
Locations (26):
- United States (18):
  - Banner Sun Health Research, Phoenix, Arizona
  - Yale University School of Medicine, New Haven, Connecticut
  - Bradenton Research Center, Bradenton, Florida
  - K2 Medical Research, Clermont, Florida
  - Advanced Clinical Research Network, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Alzheimer's Research and Treatment Center-Stuart, Stuart, Florida
  - Axiom Brain Health, Tampa, Florida
  - Charter Research, The Villages, Florida
  - Alzheimer's Research and Treatment Center, Wellington, Florida
  - Columbus Memory Center, PC, Columbus, Georgia
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - Abington Neurological Associates LTD, Abington, Pennsylvania
  - Neurology Clinic, P.C., Cordova, Tennessee
  - Kerwin Memory Center, Dallas, Texas
  - National Clinical Research-Richmond, Inc, Richmond, Virginia
- Japan (8):
  - National Center for Geriatrics and Gerontology, Ōbu, Aichi-ken
  - National Hospital Organization Hiroshima-Nishi Medical Center, Ōtake, Hiroshima
  - Keimei Memorial Hospital, Honjō, Miyazaki
  - Rijikai Medical Corporation Katayama Medical Clinic, Kurashiki, Okayama-ken
  - Tokyo Medical University Hospital, Shinjuku, Tokyo
  - Keio University Hospital, Shinjuku, Tokyo
  - Osaka Metropolitan University Hospital, Osaka
  - Yamagata Tokushukai Hospital, Yamagata

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.